CLINICAL TRIAL: NCT06969547
Title: Evaluation the Capabilities of Cardiac Mechanical Dyssynchrony in the Diagnosis of Myocardial Microvascular Dysfunction in Chronic Ischemic Heart Disease
Brief Title: Mechanical Dyssynchrony and Microvascular Dysfunction by SPECT
Acronym: MD&MD
Status: Recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Russian Science Foundation (Other)
Responsible Party: Principal Investigator, Vladimir Shipulin, Dr., Tomsk National Research Medical Center of the Russian Academy of Sciences
Other Study IDs: 249
Record Dates: First submitted 2025-04-08; First posted 2025-05-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Blood Flow Reserve; Mechanical Dyssynchrony; Coronary Arterial Disease (CAD)
Keywords: SPECT; gated MPI; mechanical dyssynchrony; dobutamine; myocardial bloow flow reserve
MeSH Terms: interventions — Blood Specimen Collection; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ischemia with no obstructive coronary arteries (INOCA): Patients with suspected chronic coronary heart disease and non-obstructive coronary artery disease according to CT coronary angiography
  Interventions: Diagnostic Test: dynamic SPECT (two-day rest/stress protocol); Diagnostic Test: gated myocardial perfusion imaging; Other: blood sampling; Diagnostic Test: Low Dose CT-scan; Diagnostic Test: CT-coronary angiography
- Obstructive coronary artery disease (CAD): Patients with chronic coronary heart disease and significant (>50%) lesion of one or more coronary artery according to CT coronary angiography
  Interventions: Diagnostic Test: dynamic SPECT (two-day rest/stress protocol); Diagnostic Test: gated myocardial perfusion imaging; Other: blood sampling; Diagnostic Test: Low Dose CT-scan; Diagnostic Test: CT-coronary angiography
- Control: Patients without evidence of coronary heart disease
  Interventions: Diagnostic Test: dynamic SPECT (two-day rest/stress protocol); Diagnostic Test: gated myocardial perfusion imaging; Other: blood sampling; Diagnostic Test: Low Dose CT-scan

INTERVENTIONS:
Diagnostic Test: dynamic SPECT (two-day rest/stress protocol) — All nuclear examinations will be performed using a hybrid specialized SPECT/CT Discovery NM/CT570C. At the first stage the passage of the bolus of the radiopharmaceutical through the chambers and the LV myocardium will be recorded at rest. Through a pre-installed intravenous catheter, a bolus of the radiopharmaceutical in a volume of 5 ml (370 MBq) will be injected at a rate of 0,5 ml/sec, after which 30 ml of saline will be injected at a rate of 2 ml/sec. Data acquisition will begin immediately before the introduction of the radiopharmaceutical. Registration of dynamic images will be performed in the "List Mode".
  At the second day stress test study will be performed (ATP at a dosage of 160 mcg/kg/min over 4 minutes). The bolus volume of the radiopharmaceutical, saline and the rate are equal to the study at rest. The time of data collection at each stage of the study will be 12 minutes. The introduction of the radiopharmaceutical will be performed at 2 minutes of the stress test.
Diagnostic Test: gated myocardial perfusion imaging — Gated MPI will be performed according to a two-day rest-stress protocol. For both stress and rest studies, the acquisition will be performed 60 minutes after the dynamic SPECT. The recording time will be 5 minutes. To correct the attenuation, a low-dose CT scan of the chest, obtained earlier with dynamic recording, will be used. The voltage on the X-ray tube will be 120 kV, the current strength will be 20 mA; tube rotation time 0.8 s; pitch 0.969:1. Radiopharmaceutical administration will be performed only once a day during dynamic SPECT.
  Immediately after recording the gMPI at rest, the patient will undergo a series of sequential injections of dobutamine at doses of 5 and 10 µg/kg/min with simultaneous recording. The duration of data collection on each dose of dobutamine will be 5 minutes.
Other: blood sampling — Indicators of:
  * endothelial dysfunction (specific endothelial cell molecule 1 (endocan, ESM1), endotelin-1)
  * severity of inflammatory response (tumor necrosis factor (TNF-α), interleukin-6 (IL-6))
  * myocardial fibrosis (matrix metalloproteinase (MMP-9)
  * myocardial dysfunction (NT-proBNP)
Diagnostic Test: Low Dose CT-scan — Scanning parameters: tube voltage 120 kV; current 435 mA; tube rotation time 0.4 s; slice thickness 2.5 mm; interslice interval 2.5 mm.
Diagnostic Test: CT-coronary angiography — The study will be performed on a 64-slice GE Discovery NM/CT 570С (GE Healthcare, Milwaukee, WI, USA) from the level of the tracheal bifurcation to the diaphragm during breath holding (6-8 s) in the prospective (for HR≤55) or retrospective (for HR>55) ECG-synchronized mode. To contrast coronary arteries, it is planned to use an intravenous infusion of 85-90 ml (at a rate of 5 ml/s) of an iodine-containing (370 mg iodine/ml) radiopaque substance.Scan will be performed with the following parameters: current strength 120 kV; voltage 300-600 mA with ECG modulation; tube rotation speed 0.4 s; pitch: 0.18-0.22 (depending on heart rate).
  Groups: Ischemia with no obstructive coronary arteries (INOCA); Obstructive coronary artery disease (CAD)

SUMMARY:
The project is aimed at studying the feasibility of mechanical dyssynchrony of the left ventricle of the heart, determined by SPECT (gated MPI), as well as its stress-induced dynamics, in the evaluation of patients with coronary microvascular dysfunction in chronic coronary heart diseasу.

DETAILED DESCRIPTION:
Each patient will have a peripheral catheter placed, blood will be drawn, followed by dynamic SPECT on a two-day rest/stress protocol, and then standard gated myocardial perfusion scintigraphy will be performed (the resting study will be followed by a study with dobutamine administration at doses of 5 and 10 µg/kg/min). The protocols will be described in detail in the Interventions section. Based on the results of dynamic SPECT, patients will be divided into 2 groups depending on the state of myocardial blood flow reserve. All nuclear examinations will be performed using a hybrid specialized SPECT/CT Discovery NM/CT570C.

1. Determination of myocardial blood flow and reserve. Myocardial blood flow and reserve will be assessed using specialized software (GE Alcyone: Dynamic Analysis Tool), two series of images will be formed from the array of primary data: 1) reflecting the passage of the radiopharmaceutical bolus through the LV cavity and myocardium from 1 to 120 seconds of the study; 2) a group of 8 dynamic tomoscintigrams (frame duration 30 s) a series of static tomoscintigrams showing the accumulation of the radiopharmaceutical in the LV walls. The next stage of data processing (bi means of of specialized software (4DM CFR) will include the analysis of static and dynamic images, with the establish of "activity-time" graphs based on areas of interest corresponding to the cavity, walls (anterior, posterior, lateral , septum and apex) and 17 segments of the polar map of the left ventricle. On the basis of the obtained graphs, indices of myocardial blood flow at rest and stress will be determined (in ml per 1 gram of tissue per minute) on the basis of which the indices of the reserve of myocardial blood flow will be determined, reflecting the MBF stress/rest ratio. These indices will be estimated for all walls, vascular regions and segments of the polar map of the left ventricle.
2. Evaluation of myocardial perfusion. To evaluate the results of myocardial perfusion, a specialized software package Corridor 4DM (University of Michigan, Ann Arbor, MI, USA) will be used with the construction of sections along the short and long axes of the heart, as well as a 17-segment polar map of the left ventricle normalized to 100%. Semi-quantitative calculation of local disorders of LV perfusion will be performed in points as follows: 0 - accumulation of radiopharmaceuticals in the myocardial segment ≥70% of the maximum; 1 - a mild decrease in accumulation (50-69%), 2 - a moderately reduced accumulation (30-49%), 3 - a pronounced decrease in accumulation (10-29%) and 4 - a severe decrease of radiopharmaceuticals accumulation (<10%). The calculation of the total violation of LV perfusion will be made as follows: a decrease <4 points will be regarded as the norm; 4-8 - as easy; 9-13 - as moderate; >13 - as a severe deterioration of myocardial perfusion. Thus, the total perfusion impairment on exercise (SSS - Summed Stress Score), at rest (SRS - Summed Rest Score), as well as SDS - Summed Difference Score - will be calculated. In addition, the indicator called transient ischemic dilatation (TID) will be determined in a specialized Quantitative Perfusion SPECT software package (QPS software, version 2013, Cedars-Sinai).
3. Evaluation of inotropic function and mechanical dyssynchrony

   To assess contractile dysfunction, we will analyze the results of gMPI obtained during dynamic acquisition with ATP (early post-exercise images), after 60 minutes after the introduction of radiopharmaceuticals, obtained with dobutamine gMPI, as well as during the study at rest. The assessment of stress-induced changes will be estimated as the difference between the score during the stress test and at rest (Δ = [value at stress] - [value at rest]). To get early post-exercise images from the array of primary data obtained during dynamic SPECT, list data from 4 to 8 will be reconstructed. The resulting images will be processed in Corridor 4DM SPECT (INVIA, Ann Arbor, MI, USA), Emory Cardiac Toolbox (Emory University/ Syntermed, Atlanta, GA), and QGS/QPS (Cedars-Sinai Medical Center, CA, USA). After construction the activity-time curve, the following parameters of the LV contractile function will be automatically estimated:

   End-systolic volume (ESV, ml); End-diastolic volume (EDV, ml); Ejection fraction (EF, %); Peak ejection rate (PER, EDV/s); Peak filling rate (PFR, EDV/s).

   After the construction of the phase histogram according to the algorithm "time to the maximum contraction", the following MD indices will be estimated automatically:

   Phase standard deviation (PSD) - standard deviation of the phase histogram; Histogram bandwidth (HBW) - phase diagram width;
4. CT coronary angiography CT coronary angiography, based on which patients will be included in the study, will be performed at the stage according to indications. The study will be conducted to assess the condition of the coronary bed on a 64-slice GE Discovery NM/CT 570C (GE Healthcare, Milwaukee, WI, USA). Unenhanced heart scans with prospective ECG synchronization and subsequent reconstruction in the 75% phase of the R-R interval will be performed to determine the coronary calcium index. The study will be conducted from the level of the tracheal bifurcation to the diaphragm. Scanning parameters will include a tube voltage of 120 kV, current of 435 mA, tube rotation time of 0.4 s, slice thickness of 2.5 mm, and an interslice interval of 2.5 mm. The coronary artery calcification index will be calculated using a dedicated Advanced Workstation (GE Healthcare) with SmartScore 4.0 software. The coronary calcium index will be determined according to the Agatston method for the trunk of the left coronary artery, the left anterior descending artery, the circumflex artery, the right coronary artery, the posterior interventricular branch, and also in total. Before starting CT coronary angiography, each patient's heart rate and blood pressure will be measured. Patients whose heart rate exceeds 65 beats per minute at the start of the study will receive an intravenous injection of 1 mg metoprolol (Betaloc, AstraZeneca). CT coronary angiography will be performed from the level of the tracheal bifurcation to the diaphragm during breath-holding (6-8 s) in prospective (for HR≤55) or retrospective (for HR>55) ECG-synchronized mode. To contrast coronary arteries, an intravenous infusion of 85-90 ml (at a rate of 5 ml/s) of an iodine-containing (370 mg iodine/ml) radiopaque substance will be used. The scan will start when a density of 200 HU is reached in the ascending aorta. CT angiography recording will be performed with the following parameters: current strength of 120 kV, voltage of 300-600 mA with ECG modulation, tube rotation speed of 0.4 s, and pitch: 0.18-0.22 (depending on heart rate). During the study, the radiation exposure will range from 1.5-3 mSv (with prospective ECG synchronization) to 15-20 mSv (with retrospective ECG synchronization). Image reconstruction will occur at the 75% phase of the cardiac cycle with a slice thickness of 0.625 mm and an interslice interval of 0.625 mm. In the presence of rhythm artifacts, images acquired with retrospective synchronization will be additionally reconstructed in the diastolic phase of the cardiac cycle (70% and 80% of the RR interval duration) and in the early diastole phase (40%, 45%, and 50% of the RR interval duration). Images with the best visualization quality of the coronary arteries will be used for further analysis. All data will be analyzed using multiplanar and curvilinear reconstructions. After the CT reconstruction, the images will be transferred and processed on a specialized workstation (AdvantageWorkstation 4.3; GE Healthcare). Segments of the coronary bed will be analyzed for the presence of atherosclerotic plaques. The quality of MSCT coronary angiograms will be assessed on a 4-point scale: 1 - excellent quality (no motion and rhythm artifacts, no significant artifacts from calcified plaques, clear identification of artery contours); 2 - good quality (minimum artifacts, minimal blurring of vessel contours); 3 - adequate quality (moderate artifacts, moderate blurring of vessels without interrupting their contours); 4 - poor quality (non-interpretable image, doubling or discontinuity of the vessel contour, lack of clear visualization of a part of the vessel). Only images with quality 1-3 will be used in the analysis. According to the American Heart Association criteria, the coronary tree will be divided into 16 segments. The degree of coronary artery stenosis will be calculated in each segment as the percentage ratio of the minimum arterial diameter at the level of the constriction to the diameter of the normal artery immediately proximal to the plaque. Stenoses ≥50% of the arterial lumen will be considered significant.
5. Epicardial adipose tissue (EAT) analysis will be performed on unenhanced images using a dedicated Advantage Workstation 4.3 (GE Healthcare). The EAT volume will be calculated in cubic millimeters automatically after manual marking of the pericardial contour in the density range from -30 to -190 HU. Also, the maximum thickness of the EJC will be measured manually on axial sections at two points: above the apex of the heart and in the right atrioventricular sulcus.

ELIGIBILITY:
Inclusion Criteria:

* Ischemia with no obstructive coronary arteries (INOCA)
* Obstructive coronary artery disease (CAD)
* Patients without evidence of coronary heart disease

Exclusion Criteria:

* Left ventricular ejection fraction <55% according to echocardiography;
* History of myocardial infarction/revascularization;
* hypertension: systolic blood pressure >180 mm Hg. Art., diastolic BP>110 mm Hg. Art.;
* systolic arterial hypotension <80 mm Hg. Art.;
* atrial fibrillation;
* AV blockade of the III degree; sick sinus syndrome;
* massive pulmonary embolism (PE) with a high degree of pulmonary hypertension;
* the presence of significant valvular pathology (mitral insufficiency ≥ 3 degrees, aortic insufficiency ≥ 3 degrees, tricuspid regurgitation ≥ 3 degrees).
* severe course of bronchial asthma, chronic obstructive pulmonary disease;
* decompensated type 2 diabetes,
* severe liver or kidney failure (glomerular filtration rate <50 ml/min/1.73 m3 (CKD-EPI),
* morbid obesity (body mass index >45);
* history of myocarditis
* indications of poor drug tolerance;
* oncological diseases;
* chronic alcoholism, mental disorders;
* other severe comorbidity,
* refusal to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Tomsk, Russia
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Decreased myocardial blood flow reserve | 1 day
  Baseline decrease in myocardial blood flow reserve according to dynamic SPECT <2.0

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Shipulin, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Tomsk NRMC Cardiology Research Institute, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No